CLINICAL TRIAL: NCT02234843
Title: Multicenter, Open-label, Active-controlled, Randomized Study to Evaluate the Efficacy and Safety of an age-and Body Weight-adjusted Rivaroxaban Regimen Compared to Standard of Care in Children With Acute Venous Thromboembolism
Brief Title: EINSTEIN Junior: Oral Rivaroxaban in Children With Venous Thrombosis
Acronym: EINSTEIN Jr
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14372; 2014-000565-47 (EudraCT Number)
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Results first posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Venous Thromboembolism
Keywords: Pediatric
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BAY59-7939 (Experimental): Rivaroxaban (tablets and oral suspension) Dose: Age and body weight-adjusted dosing of rivaroxaban to achieve a similar exposure as that observed in adults treated for venous thromboembolism (VTE) with 20 mg rivaroxaban.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Standard of Care (Experimental): Subcutaneous low molecular weight heparin (LMWH), subcutaneous fondaparinux and/or oral vitamin K antagonist (VKA) Dose : as per standard of care
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Age and body weight-adjusted dosing equivalent to 20 mg rivaroxaban in adults, once daily or twice daily, as tablets
  Arms: BAY59-7939
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Age and body weight-adjusted dosing equivalent to 20 mg rivaroxaban in adults, once daily, twice daily or three times daily, as oral suspension
  Arms: BAY59-7939
Drug: Standard of Care — LMWH (low molecular weight heparin) or fondaparinux or vitamin K antagonist (VKA) therapy.
  dose : as per standard of care
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate comparative efficacy and safety of rivaroxaban to standard of care in children with acute venous thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Children aged birth to < 18 years with confirmed venous thromboembolism who receive initial treatment with therapeutic dosages of UFH (unfractionated heparin), LMWH (low molecular weight heparin) or fondaparinux and require anticoagulant therapy for at least 90 days. However, children aged birth to < 2 years with catheter-related thrombosis require anticoagulant therapy for at least 30 days.
* For children younger than 6 months:

  * Gestational age at birth of at least 37 weeks.
  * Oral feeding/nasogastric/gastric feeding for at least 10 days.
  * Body weight ≥2600 g

Exclusion Criteria:

* Active bleeding or bleeding risk contraindicating anticoagulant therapy
* An estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m*2 (in children younger than 1 year, serum creatinine results above 97.5th percentile excludes participation)
* Hepatic disease which is associated with either: coagulopathy leading to a clinically relevant bleeding risk, or ALT> 5x upper level of normal (ULN) or total bilirubin > 2x ULN with direct bilirubin > 20% of the total
* Platelet count < 50 x 109/L
* Sustained uncontrolled hypertension defined as > 95th age percentile
* Life expectancy < 3 months
* Concomitant use of strong inhibitors of both cytochrome P450 isoenzyme 3A4 (CYP3A4) and P-glycoprotein (P-gp), including but not limited to all human immunodeficiency virus protease inhibitors and the following azole antimycotics agents: ketoconazole, itraconazole, voriconazole, posaconazole, if used systemically
* Concomitant use of strong inducers of CYP3A4, including but not limited to rifampicin, rifabutin, phenobarbital, phenytoin and carbamazepine
* Childbearing potential without proper contraceptive measures, pregnancy or breast feeding

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (103):
- United States (22):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - San Diego, California
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Pensacola, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lansing, Michigan
  - Kansas City, Missouri
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
- San Miguel de Tucumán, Tucumán Province, Argentina
- Australia (2):
  - Parkville, Victoria
  - South Brisbane
- Austria (4):
  - Graz, Styria
  - Innsbruck, Tyrol
  - Linz, Upper Austria
  - Vienna
- Belgium (3):
  - Bruxelles - Brussel
  - Edegem
  - Leuven
- Brazil (3):
  - Campinas, São Paulo
  - São Paulo, São Paulo
  - São Paulo
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- China (3):
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
- Turku, Finland
- France (3):
  - Montpellier
  - Paris
  - Toulouse
- Germany (4):
  - Erlangen, Bavaria
  - Dresden, Saxony
  - Halle, Saxony-Anhalt
  - Berlin
- Hong Kong, Hong Kong
- Budapest, Hungary
- Crumlin, Dublin, Ireland
- Israel (4):
  - Afula
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
- Italy (3):
  - Milan, Lombardy
  - Turin, Piedmont
  - Padua, Veneto
- Japan (3):
  - Ōbu, Aichi-ken
  - Azumino, Nagano
  - Bunkyo-ku, Tokyo
- Mexico (2):
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
- Netherlands (5):
  - Amsterdam
  - Groningen
  - Nijmegen
  - Rotterdam
  - Utrecht
- Carnaxide, Lisbon District, Portugal
- Russia (8):
  - Kazan'
  - Kemerovo
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Volgograd
  - Yekaterinburg
- Singapore, Singapore
- Bratislava, Slovakia
- Spain (3):
  - Esplugues de Llobregat, Barcelona
  - A Coruña
  - Barcelona
- Solna, Sweden
- Switzerland (3):
  - Bern
  - Lucerne
  - Zurich
- Turkey (Türkiye) (3):
  - Adana
  - Istanbul
  - Konya
- United Kingdom (10):
  - Newcastle upon Tyne, Tyne and Wear
  - Birmingham, West Midlands
  - Leeds, West Yorkshire
  - Cardiff
  - Edinburgh
  - Glasgow
  - London
  - Manchester
  - Oxford
  - Sheffield

REFERENCES:
- [Derived] Palumbo JS, Lensing AWA, Brandao LR, Hooimeijer HL, Kenet G, van Ommen H, Pap AF, Majumder M, Kubitza D, Thelen K, Willmann S, Prins MH, Monagle P, Male C. Anticoagulation in pediatric cancer-associated venous thromboembolism: a subgroup analysis of EINSTEIN-Jr. Blood Adv. 2022 Nov 22;6(22):5821-5828. doi: 10.1182/bloodadvances.2022008160. PMID 36006613
- [Derived] Connor P, Sanchez van Kammen M, Lensing AWA, Chalmers E, Kallay K, Hege K, Simioni P, Biss T, Bajolle F, Bonnet D, Grunt S, Kumar R, Lvova O, Bhat R, Van Damme A, Palumbo J, Santamaria A, Saracco P, Payne J, Baird S, Godder K, Labarque V, Male C, Martinelli I, Morales Soto M, Motwani J, Shah S, Hooimeijer HL, Prins MH, Kubitza D, Smith WT, Berkowitz SD, Pap AF, Majumder M, Monagle P, Coutinho JM. Safety and efficacy of rivaroxaban in pediatric cerebral venous thrombosis (EINSTEIN-Jr CVT). Blood Adv. 2020 Dec 22;4(24):6250-6258. doi: 10.1182/bloodadvances.2020003244. PMID 33351120
- [Derived] Thom K, Lensing AWA, Nurmeev I, Bajolle F, Bonnet D, Kenet G, Massicotte MP, Karakas Z, Palumbo JS, Saracco P, Amedro P, Chain J, Chan AK, Ikeyama T, Lam JCM, Gauger C, Pap AF, Majumder M, Kubitza D, Smith WT, Berkowitz SD, Prins MH, Monagle P, Young G, Male C. Safety and efficacy of anticoagulant therapy in pediatric catheter-related venous thrombosis (EINSTEIN-Jr CVC-VTE). Blood Adv. 2020 Oct 13;4(19):4632-4639. doi: 10.1182/bloodadvances.2020002637. PMID 33002131
- [Derived] Male C, Lensing AWA, Palumbo JS, Kumar R, Nurmeev I, Hege K, Bonnet D, Connor P, Hooimeijer HL, Torres M, Chan AKC, Kenet G, Holzhauer S, Santamaria A, Amedro P, Chalmers E, Simioni P, Bhat RV, Yee DL, Lvova O, Beyer-Westendorf J, Biss TT, Martinelli I, Saracco P, Peters M, Kallay K, Gauger CA, Massicotte MP, Young G, Pap AF, Majumder M, Smith WT, Heubach JF, Berkowitz SD, Thelen K, Kubitza D, Crowther M, Prins MH, Monagle P; EINSTEIN-Jr Phase 3 Investigators. Rivaroxaban compared with standard anticoagulants for the treatment of acute venous thromboembolism in children: a randomised, controlled, phase 3 trial. Lancet Haematol. 2020 Jan;7(1):e18-e27. doi: 10.1016/S2352-3026(19)30219-4. Epub 2019 Nov 5. PMID 31699660
- [Derived] Monagle P, Lensing AWA, Thelen K, Martinelli I, Male C, Santamaria A, Samochatova E, Kumar R, Holzhauer S, Saracco P, Simioni P, Robertson J, Grangl G, Halton J, Connor P, Young G, Molinari AC, Nowak-Gottl U, Kenet G, Kapsa S, Willmann S, Pap AF, Becka M, Twomey T, Beyer-Westendorf J, Prins MH, Kubitza D; EINSTEIN-Jr Phase 2 Investigators. Bodyweight-adjusted rivaroxaban for children with venous thromboembolism (EINSTEIN-Jr): results from three multicentre, single-arm, phase 2 studies. Lancet Haematol. 2019 Oct;6(10):e500-e509. doi: 10.1016/S2352-3026(19)30161-9. Epub 2019 Aug 13. PMID 31420317
- [Derived] Lensing AWA, Male C, Young G, Kubitza D, Kenet G, Patricia Massicotte M, Chan A, Molinari AC, Nowak-Goettl U, Pap AF, Adalbo I, Smith WT, Mason A, Thelen K, Berkowitz SD, Crowther M, Schmidt S, Price V, Prins MH, Monagle P. Rivaroxaban versus standard anticoagulation for acute venous thromboembolism in childhood. Design of the EINSTEIN-Jr phase III study. Thromb J. 2018 Dec 21;16:34. doi: 10.1186/s12959-018-0188-y. eCollection 2018. PMID 30598642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 109 study centers in 28 countries: Argentina, Australia, Austria, Belgium, Brazil, Canada, China, Finland, France, Germany, Hong Kong, Hungary, Ireland, Israel, Italy, Japan, Mexico, Netherlands, Portugal, Russia, Singapore, Slovakia, Spain, Sweden, Switzerland, Turkey, UK, and USA between 13 Nov 2014 and 30 Jan 2019.
Pre-assignment Details: A total of 520 children were screened for this study. Twenty children did not pass the screen of inclusion/exclusion criteria. A total of 500 children were randomized 2:1 to study treatment.
Groups:
- Rivaroxaban, Aged 12-<18: Children aged 12-<18 years randomized to rivaroxaban received either tablet or oral suspension after at least 5 days administration of initial therapy with UFH/LMWH/fondaparinux . Children with body weight of ≥ 20 kg received rivaroxaban tablets or oral suspension.
- Rivaroxaban, Aged 6-<12: Children aged 6-<12 years randomized to rivaroxaban received either tablet or oral suspension after at least 5 days administration of initial therapy with UFH/LMWH/fondaparinux . Children with body weight of ≥ 20 kg received rivaroxaban tablets or oral suspension. Children with body weight of < 20 kg received rivaroxaban as oral suspension.
- Rivaroxaban, Aged 2-<6: Children aged 2-<6 years randomized to rivaroxaban received oral suspension after at least 5 days administration of initial therapy with UFH/LMWH/fondaparinux . Children with body weight of ≥ 20 kg received rivaroxaban tablets or oral suspension. Children with body weight of < 20 kg received rivaroxaban as oral suspension.
- Rivaroxaban, Aged 0.5-<2: Children aged 0.5-<2 years randomized to rivaroxaban received oral suspension after at least 5 days administration of initial therapy with UFH/LMWH/fondaparinux . Children with body weight of < 20 kg received rivaroxaban as oral suspension.
- Rivaroxaban, Aged Birth-<0.5: Children aged birth-<0.5 years randomized to rivaroxaban received oral suspension after at least 5 days administration of initial therapy with UFH/LMWH/fondaparinux . Children with body weight of < 20 kg received rivaroxaban as oral suspension.
- Comparator, Aged 12-<18: Children aged 12-<18 years randomized to the comparator group continued with unfractionated heparin (UFH), low molecular weight heparin (LMWH) or fondaparinux or may switch to Vitamin K Antagonist (VKA) therapy. VKA dosages were adjusted to maintain the international normalized ratio (INR) within the therapeutic range (target 2.5, range 2.0 - 3.0). UFH, LMWH or fondaparinux could be discontinued once the INR was above 2.0 on two separate occasions, 24 hours apart.
- Comparator, Aged 6-<12: Children aged 6-<12 years randomized to the comparator group continued with unfractionated heparin (UFH), low molecular weight heparin (LMWH) or fondaparinux or may switch to VKA therapy. VKA dosages were adjusted to maintain the INR within the therapeutic range (target 2.5, range 2.0 - 3.0). UFH, LMWH or fondaparinux could be discontinued once the INR was above 2.0 on two separate occasions, 24 hours apart.
- Comparator, Aged 2-<6: Children aged 2-<6 years randomized to the comparator group continued with unfractionated heparin (UFH), low molecular weight heparin (LMWH) or fondaparinux or may switch to VKA therapy. VKA dosages were adjusted to maintain the INR within the therapeutic range (target 2.5, range 2.0 - 3.0). UFH, LMWH or fondaparinux could be discontinued once the INR was above 2.0 on two separate occasions, 24 hours apart.
- Comparator, Aged 0.5-<2: Children aged 0.5-<2 years randomized to the comparator group continued with unfractionated heparin (UFH), low molecular weight heparin (LMWH) or fondaparinux or may switch to VKA therapy. VKA dosages were adjusted to maintain the INR within the therapeutic range (target 2.5, range 2.0 - 3.0). UFH, LMWH or fondaparinux could be discontinued once the INR was above 2.0 on two separate occasions, 24 hours apart.
- Comparator, Aged Birth-<0.5: Children aged birth-<0.5 years randomized to the comparator group continued with unfractionated heparin (UFH), low molecular weight heparin (LMWH) or fondaparinux or may switch to VKA therapy. VKA dosages were adjusted to maintain the INR within the therapeutic range (target 2.5, range 2.0 - 3.0). UFH, LMWH or fondaparinux could be discontinued once the INR was above 2.0 on two separate occasions, 24 hours apart.
Period: Overall Study
Arm/Group | Rivaroxaban, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5 | Comparator, Aged 12-<18 | Comparator, Aged 6-<12 | Comparator, Aged 2-<6 | Comparator, Aged 0.5-<2 | Comparator, Aged Birth-<0.5
Started | 184 | 67 | 47 | 21 | 16 | 92 | 34 | 22 | 9 | 8
Completed | 162 | 61 | 44 | 16 | 14 | 79 | 32 | 20 | 8 | 8
Not Completed | 22 | 6 | 3 | 5 | 2 | 13 | 2 | 2 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Efficacy outcome reached | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Patient convenience | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 1 | 0 | 0 | 7 | 0 | 0 | 0 | 0
Not completed — Recovery | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 5 | 1 | 1 | 3 | 2 | 1 | 0 | 0 | 1 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Comparator, Aged 12-<18: Children aged 12-<18 years randomized to the comparator group continued with unfractionated heparin (UFH), low molecular weight heparin (LMWH) or fondaparinux or may switch to VKA therapy. VKA dosages were adjusted to maintain the INR within the therapeutic range (target 2.5, range 2.0 - 3.0). UFH, LMWH or fondaparinux could be discontinued once the INR was above 2.0 on two separate occasions, 24 hours apart.
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5 | Comparator, Aged 12-<18 | Comparator, Aged 6-<12 | Comparator, Aged 2-<6 | Comparator, Aged 0.5-<2 | Comparator, Aged Birth-<0.5 | Total
Number analyzed (Participants) | 184 | 67 | 47 | 21 | 16 | 92 | 34 | 22 | 9 | 8 | 500
Age, Customized [Count of Participants; unit: Participants]
  12-<18 years | 184 | 0 | 0 | 0 | 0 | 92 | 0 | 0 | 0 | 0 | 276
  6-<12 years | 0 | 67 | 0 | 0 | 0 | 0 | 34 | 0 | 0 | 0 | 101
  2-<6 years | 0 | 0 | 47 | 0 | 0 | 0 | 0 | 22 | 0 | 0 | 69
  0.5-<2 years | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 9 | 0 | 30
  Birth-<0.5 years | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 8 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 24 | 24 | 10 | 5 | 55 | 15 | 9 | 5 | 1 | 245
  Male | 87 | 43 | 23 | 11 | 11 | 37 | 19 | 13 | 4 | 7 | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 164 | 58 | 42 | 15 | 12 | 79 | 26 | 19 | 8 | 6 | 429
  Not Hispanic or Latino | 7 | 5 | 1 | 3 | 1 | 6 | 5 | 1 | 0 | 0 | 29
  Unknown or Not Reported | 13 | 4 | 4 | 3 | 3 | 7 | 3 | 2 | 1 | 2 | 42

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rates of All Symptomatic Recurrent Venous Thromboembolism During the Main Treatment Period
Description: The Central independent adjudication committee (CIAC) classified symptomatic recurrent venous thromboembolism (VTE). Incidence = number of events / number at risk, where: number of events = number of subjects having the event in the time window. number at risk = number of subjects in reference population
Time Frame: During the main study treatment period (i.e., 3 months, except for children with central venous catheter venous thromboembolism (CVC-VTE) aged <2 years for whom it was 1 month)
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Rivaroxaban Group: Children randomized to rivaroxaban received either tablet or oral suspension after at least 5 days administration of initial therapy with UFH/LMWH/fondaparinux. Children with body weight of ≥ 20 kg received rivaroxaban tablets or oral suspension. Children with body weight of < 20 kg received rivaroxaban as oral suspension.
- Comparator Group: Children randomized to the comparator group will continue with UFH, LMWH or fondaparinux or may switch to VKA therapy. VKA dosages will be adjusted to maintain the INR within the therapeutic range (target 2.5, range 2.0 - 3.0). UFH, LMWH or fondaparinux can be discontinued once the INR is above 2.0 on two separate occasions, 24 hours apart
Arm/Group | Rivaroxaban Group | Comparator Group
Number analyzed (Participants) | 335 | 165
Percentage of participants | 1.2 [0.4 to 3.0] | 3.0 [1.2 to 6.6]
Statistical Analysis 1: Comparison: Rivaroxaban Group vs Comparator Group; Test type: Other; p = 0.1509, Expl. Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.11 to 1.41]

2. Primary Outcome: Incidence Rates of All Symptomatic Recurrent Venous Thromboembolism During the Main Treatment Period
Description: as for outcome 1
Time Frame: During the main study treatment period (i.e., 3 months, except for children with CVC-VTE aged <2 years for whom it was 1 month)
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivaroxaban, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5 | Comparator, Aged 12-<18 | Comparator, Aged 6-<12 | Comparator, Aged 2-<6 | Comparator, Aged 0.5-<2 | Comparator, Aged Birth-<0.5
Number analyzed (Participants) | 184 | 67 | 47 | 21 | 16 | 92 | 34 | 22 | 9 | 8
Percentage of participants | 2.2 (0.7) [0.7 to 5.3] | 0.0 (0.0) [0.0 to 5.3] | 0.0 (0.0) [0.0 to 6.8] | 0.0 (0.0) [0.0 to 8.3] | 0.0 (0.0) [0.0 to 14.6] | 3.3 (0.9) [0.9 to 8.6] | 2.9 (0.2) [0.2 to 15.1] | 4.5 (0.2) [0.2 to 20.7] | 0.0 (0.0) [0.0 to 18.4] | 0.0 (0.0) [0.0 to 29.9]

3. Primary Outcome: Incidence Rates of All Symptomatic Recurrent Venous Thromboembolism During Extended Treatment Period
Description: Incidence rates for all children except those aged < 2 years with catheter-related thrombosis. If no participant in the specific subgroup entered in the specific optional extension period, no analysis of an outcome was possible., The Central independent adjudication committee (CIAC) classified symptomatic recurrent venous thromboembolism (VTE). Incidence = number of events / number at risk, where: number of events = number of subjects having the event in the time window. number at risk = number of subjects in reference Population.
Time Frame: During extended treatment period: up to month 12.
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivaroxaban, Aged 12-<18 | Comparator, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5 | Comparator, Aged 6-<12 | Comparator, Aged 2-<6 | Comparator, Aged 0.5-<2 | Comparator, Aged Birth-<0.5
Number analyzed (Participants) | 93 | 46 | 21 | 19 | 0 | 2 | 8 | 7 | 1 | 1
Percentage of participants
  Extension 1 (month 3 to 6) | 0.0 [0.0 to 3.8] | 2.2 [0.1 to 10.9] | 0.0 [0.0 to 14.6] | 0.0 [0.0 to 16.3] |  | 0.0 [0.0 to 77.6] | 0.0 [0.0 to 14.6] | 0.0 [0.0 to 37.7] | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 95.0]
  Extension 2 (month 6 to 9): number analyzed (Participants) | 38 | 19 | 9 | 6 | 0 | 0 | 3 | 3 | 0 | 0
  Extension 2 (month 6 to 9) | 2.6 [0.1 to 13.4] | 5.3 [0.3 to 24.4] | 0.0 [0.0 to 29.9] | 0.0 [0.0 to 40.2] |  |  | 0.0 [0.0 to 63.2] | 0.0 [0.0 to 77.6] |  |
  Extension 3 (month 9 to 12): number analyzed (Participants) | 26 | 14 | 3 | 2 | 0 | 0 | 1 | 2 | 0 | 0
  Extension 3 (month 9 to 12) | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 23.0] | 0.0 [0.0 to 63.2] | 0.0 [0.0 to 77.6] |  |  | 0.0 [0.0 to 95.2] | 0.0 [0.0 to 77.6] |  |

4. Primary Outcome: Number of Subjects With the Composite of All Symptomatic Recurrent Venous Thromboembolism During the 30 Days Post-study Treatment Period (i.e. >2 and ≤ 30 Days After Stop of Study Medication)
Description: The Central independent adjudication committee (CIAC) classified symptomatic recurrent venous thromboembolism (VTE). Age group with primary efficacy outcome was reported.
Time Frame: More than 2 and up to 30 days after stop of study medication
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban, Aged 12-<18 | Comparator, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5 | Comparator, Aged 6-<12 | Comparator, Aged 2-<6 | Comparator, Aged 0.5-<2 | Comparator, Aged Birth-<0.5
Number analyzed (Participants) | 184 | 92 | 67 | 47 | 21 | 16 | 34 | 22 | 9 | 8
Participants | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Incidence Rates of the Composite of Treatment Emergent Overt Major Bleeding and Clinically Relevant Non-major (CRNM) Bleeding During Main Treatment Period
Description: The Central independent adjudication committee (CIAC) classified bleeding as: Major bleeding defined as overt bleeding and: · associated with a fall in hemoglobin of 2 g/dL or more, or leading to a transfusion of the equivalent of 2 or more units of packed red blood cells or whole blood in adults, or occurring in a critical site, e.g. intracranial, intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, retroperitoneal, or contributing to death. Clinically relevant non-major bleeding defined as overt bleeding not meeting the criteria for major bleeding, but associated with: medical intervention, or unscheduled contact (visit or telephone call) with a physician, or (temporary) cessation of study treatment, or discomfort for the child such as pain or impairment of activities of daily life (such as loss of school days or hospitalization).
Time Frame: as for outcome 2
Population: Safety analysis set (SAF)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivaroxaban Group | Comparator Group
Number analyzed (Participants) | 329 | 162
Percentage of participants | 3 [1.6 to 5.5] | 1.9 [0.5 to 3.3]

6. Primary Outcome: Incidence Rates of the Composite of Treatment Emergent Overt Major Bleeding and Clinically Relevant Non-major (CRNM) Bleeding During Main Treatment Period
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Safety analysis set (SAF)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivaroxaban, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5 | Comparator, Aged 12-<18 | Comparator, Aged 6-<12 | Comparator, Aged 2-<6 | Comparator, Aged 0.5-<2 | Comparator, Aged Birth-<0.5
Number analyzed (Participants) | 180 | 67 | 46 | 21 | 15 | 89 | 34 | 22 | 9 | 8
Percentage of participants | 1.7 (0.5) [0.5 to 4.7] | 3.0 (0.5) [0.5 to 9.6] | 6.5 (1.8) [1.8 to 17.7] | 4.8 (0.2) [0.2 to 21.8] | 6.7 (0.3) [0.3 to 30.2] | 2.2 (0.4) [0.4 to 7.3] | 0.0 (0.0) [0.0 to 9.0] | 0.0 (0.0) [0.0 to 13.9] | 11.1 (0.6) [0.6 to 44.3] | 0.0 (0.0) [0.0 to 34.9]

7. Primary Outcome: Incidence Rates of the Composite of Treatment Emergent Overt Major Bleeding and Clinically Relevant Non-major (CRNM) Bleeding During Extended Treatment Period
Description: Incidence rates for all children except those aged < 2 years with catheter-related thrombosis. If no participant entered in the specific optional extension period, no analysis of an outcome was possible. The CIAC classified bleeding as: Major bleeding defined as overt bleeding and: associated with a fall in hemoglobin of 2 g/dL or more, or leading to a transfusion of the equivalent of 2 or more units of packed red blood cells or whole blood in adults, or occurring in a critical site, e.g. intracranial, intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, retroperitoneal, or contributing to death. Clinically relevant non-major bleeding defined as overt bleeding not meeting the criteria for major bleeding, but associated with: medical intervention, or unscheduled contact with a physician, or (temporary) cessation of study treatment, or discomfort for the child such as pain or impairment of activities of daily life.
Time Frame: During extended treatment period: up to month 12.
Population: Safety analysis set (SAF)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivaroxaban, Aged 12-<18 | Rivaroxaban, Aged 0.5-<2 | Comparator, Aged 12-<18 | Comparator, Aged 0.5-<2 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged Birth-<0.5 | Comparator, Aged 6-<12 | Comparator, Aged 2-<6 | Comparator, Aged Birth-<0.5
Number analyzed (Participants) | 93 | 0 | 46 | 1 | 21 | 19 | 2 | 8 | 7 | 1
Percentage of participants
  Extension 1 (month 3 to 6) | 1.1 [0.1 to 5.3] |  | 0.0 [0.0 to 6.9] | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 14.6] | 0.0 [0.0 to 16.3] | 0.0 [0.0 to 77.6] | 0.0 [0.0 to 34.9] | 0.0 [0.0 to 37.7] | 0.0 [0.0 to 95.0]
  Extension 2 (month 6 to 9): number analyzed (Participants) | 38 | 0 | 19 | 0 | 9 | 6 | 0 | 3 | 2 | 0
  Extension 2 (month 6 to 9) | 2.6 [0.1 to 13.4] |  | 5.3 [0.3 to 24.4] |  | 0.0 [0.0 to 29.9] | 0.0 [0.0 to 40.2] |  | 0.0 [0.0 to 63.2] | 0.0 [0.0 to 77.6] |
  Extension 3 (month 9 to 12): number analyzed (Participants) | 26 | 0 | 46 | 0 | 3 | 2 | 0 | 1 | 2 | 0
  Extension 3 (month 9 to 12) | 0.0 [0.0 to 11.6] |  | 0.0 [0.0 to 23.0] |  | 0.0 [0.0 to 63.2] | 0.0 [0.0 to 77.6] |  | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 77.6] |

8. Secondary Outcome: Incidence Rates of the Composite of All Symptomatic Recurrent Venous Thromboembolism and Asymptomatic Deterioration in Thrombotic Burden on Repeat Imaging During the Main Treatment Period
Description: The secondary efficacy outcome defined as the composite of all symptomatic recurrent venous thromboembolism and asymptomatic deterioration on repeat imaging as assessed by central independent adjudication committee. (CIAC) Incidence = number of events / number at risk, where: number of events = number of subjects having the event in the time window. number at risk = number of subjects in reference population
Time Frame: as for outcome 2
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivaroxaban, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5 | Comparator, Aged 12-<18 | Comparator, Aged 6-<12 | Comparator, Aged 2-<6 | Comparator, Aged 0.5-<2 | Comparator, Aged Birth-<0.5
Number analyzed (Participants) | 184 | 67 | 47 | 21 | 16 | 92 | 34 | 22 | 9 | 8
Percentage of participants | 2.2 (0.7) [0.7 to 5.3] | 0.0 (0.0) [0.0 to 5.3] | 2.1 (0.1) [0.1 to 10.7] | 0.0 (0.0) [0.0 to 14.6] | 0.0 (0.0) [0.0 to 19.8] | 4.3 (1.5) [1.5 to 10.3] | 2.9 (0.2) [0.2 to 15.1] | 4.5 (0.2) [0.2 to 20.7] | 0.0 (0.0) [0.0 to 29.9] | 0.0 (0.0) [0.0 to 34.9]

9. Secondary Outcome: AUC(0-24)ss in Plasma
Description: AUC(0-24)ss: Area under the concentration vs. time curve from time 0 to 24 hours at steady state.
Time Frame: over 24 hours
Population: Pharmacokinetics analysis set (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per liter
Arm/Group | Rivaroxaban, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5
Number analyzed (Participants) | 173 | 65 | 44 | 21 | 13
microgram*hour per liter | 2120 (26.4) [lower limit 26.4] | 1960 (31.7) [lower limit 31.7] | 2380 (40.7) [lower limit 40.7] | 1840 (36.4) [lower limit 36.4] | 1590 (29.6) [lower limit 29.6]

10. Secondary Outcome: Cmax,ss in Plasma
Description: Maximum drug concentration in measured matrix at steady state during a dosage interval
Time Frame: 0 hours to 24 hours, 0 hours to 12 hours or 0 hours to 8 hours (one dosing interval in steady state)
Population: Pharmacokinetics analysis set (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter
Arm/Group | Rivaroxaban, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5
Number analyzed (Participants) | 173 | 65 | 44 | 21 | 13
microgram per liter | 237 (20.6) [lower limit 20.6] | 184 (36.2) [lower limit 36.2] | 182 (31.2) [lower limit 31.2] | 136 (29.4) [lower limit 29.4] | 119 (24.1) [lower limit 24.1]

11. Secondary Outcome: Ctrough,ss in Plasma
Description: Ctrough,ss refers to the drug concentration at the end of the dosage interval at steady state
Time Frame: 0 hours to 24 hours, 0 hours to 12 hours or 0 hours to 8 hours(one sampling interval in steady state)
Population: Pharmacokinetics analysis set (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter
Arm/Group | Rivaroxaban, Aged 12-<18 | Rivaroxaban, Aged 6-<12 | Rivaroxaban, Aged 2-<6 | Rivaroxaban, Aged 0.5-<2 | Rivaroxaban, Aged Birth-<0.5
Number analyzed (Participants) | 173 | 65 | 44 | 21 | 13
microgram per liter | 20.7 (45.8) [lower limit 45.8] | 21.4 (62.7) [lower limit 62.7] | 31.6 (70.1) [lower limit 70.1] | 22.9 (68.6) [lower limit 68.6] | 18.5 (50.4) [lower limit 50.4]

12. Secondary Outcome: Prothrombin Time (PT) Ratios to Baseline: Rivaroxaban Administered Once Daily (Suspension and Tablet) in the Age Group 12-<18 Years
Description: Prothrombin time (PT) is a global clotting test assessing the extrinsic pathway of the blood coagulation cascade. The test is sensitive for deficiencies of Factors II, V, VII, and X, with sensitivity being best for Factors V, VII, and X and less pronounced for Factor II. The initial read-out is in seconds.
Time Frame: Up to 4 hours post dose on Day30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 12-<18
Number analyzed (Participants) | 156
ratio
  Day 30 (0.5-1.5h) n=156 | 1.29 (0.28)
  Day 30 (2.5-4h) n=150: number analyzed (Participants) | 150
  Day 30 (2.5-4h) n=150 | 1.57 (0.36)
  Day 60 (2-8h) n=156 | 1.52 (0.29)

13. Secondary Outcome: Prothrombin Time (PT) Ratios to Baseline: Rivaroxaban Administered Once Daily (Suspension and Tablet) in the Age Group 6-<12 Years
Description: as for outcome 12
Time Frame: Up to 4 hours post dose on Day30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 6-<12
Number analyzed (Participants) | 20
ratio
  Day 30 (0.5-1.5h) n=18: number analyzed (Participants) | 18
  Day 30 (0.5-1.5h) n=18 | 1.46 (0.25)
  Day 30 (2.5-4h) n=20 | 1.67 (0.39)
  Day 60 (2-8h) n=20 | 1.52 (0.33)

14. Secondary Outcome: Prothrombin Time (PT) Ratios to Baseline: Rivaroxaban Administered Twice Daily (Suspension and Tablet) in the Age Group 6-<12 Years
Description: as for outcome 12
Time Frame: Up to 4 hours post dose on Day30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 6-<12
Number analyzed (Participants) | 34
ratio
  Day 30 (0.5-1.5h) n=33: number analyzed (Participants) | 33
  Day 30 (0.5-1.5h) n=33 | 1.17 (0.23)
  Day 30 (2.5-4h) n=33: number analyzed (Participants) | 33
  Day 30 (2.5-4h) n=33 | 1.26 (0.22)
  Day 60 (2-8h) n=34 | 1.21 (0.19)

15. Secondary Outcome: Prothrombin Time (PT) Ratios to Baseline: Rivaroxaban Administered Twice Daily (Suspension) in the Age Group 2-<6 Years
Description: Prothrombin time (PT) is a global clotting test assessing the extrinsic pathway of the blood coagulation cascade. The test is sensitive for deficiencies of Factors II, V, VII, and X, with sensitivity being best for Factors V, VII, and X and less pronounced for Factor II. The initial read-out is in seconds. 'NA' denotes the data that cannot be calculated.
Time Frame: Up to 4 hours post dose on Day30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 2-<6
Number analyzed (Participants) | 34
ratio
  Day 30 (0.5-1.5h) n=1: number analyzed (Participants) | 1
  Day 30 (0.5-1.5h) n=1 | 0.99 (NA) — 'NA' denotes data that cannot be calculated.
  Day 30 (2.5-4h) n=34 | 1.36 (0.28)
  Day 60 (2-8h) n=32: number analyzed (Participants) | 32
  Day 60 (2-8h) n=32 | 1.33 (0.26)

16. Secondary Outcome: Prothrombin Time (PT) Ratios to Baseline: Rivaroxaban Administered Twice Daily (Suspension) in the Age Group 0.5-<2 Years
Description: as for outcome 15
Time Frame: Up to 4 hours post dose on Day30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 0.5-<2
Number analyzed (Participants) | 2
ratio
  Day 30 (0.5-1.5h) n=0: number analyzed (Participants) | 0
  Day 30 (2.5-4h) n=1: number analyzed (Participants) | 1
  Day 30 (2.5-4h) n=1 | 1.41 (NA) — 'NA' denotes data that cannot be calculated.
  Day 60 (2-8h) n=2 | 1.05 (0.17)

17. Secondary Outcome: Prothrombin Time (PT) Ratios to Baseline: Rivaroxaban Administered Three Times Daily (Suspension) in the Age Group 2-<6 Years
Description: as for outcome 12
Time Frame: Up to 3 hours post dose on Day30, and up to 6 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 2-<6
Number analyzed (Participants) | 4
ratio
  Day 30 (0.5-3h) n=4 | 1.87 (1.09) [lower limit 1.09]
  Day 60 (2-6h) n=4 | 1.32 (0.12) [lower limit 0.12]

18. Secondary Outcome: Prothrombin Time (PT) Ratios to Baseline: Rivaroxaban Administered Three Times Daily (Suspension) in the Age Group 0.5-<2 Years
Description: as for outcome 12
Time Frame: Up to 3 hours post dose on Day30, and up to 6 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratios
Arm/Group | Rivaroxaban, Aged 0.5-<2
Number analyzed (Participants) | 9
ratios
  Day 30 (0.5-3h) n=9 | 1.25 (0.18)
  Day 60 (2-6h) n=7: number analyzed (Participants) | 7
  Day 60 (2-6h) n=7 | 2.00 (2.22)

19. Secondary Outcome: Prothrombin Time (PT) Ratios to Baseline: Rivaroxaban Administered Three Times Daily (Suspension) in the Age Group Birth-<0.5 Years
Description: as for outcome 12
Time Frame: Up to 3 hours post dose on Day30, and up to 6 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged Birth-<0.5
Number analyzed (Participants) | 11
ratio
  Day 30 (0.5-3h) n=11 | 1.35 (0.20)
  Day 60 (2-6h) n=4: number analyzed (Participants) | 4
  Day 60 (2-6h) n=4 | 1.45 (0.16)

20. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Ratios to Baseline: Rivaroxaban Administered Once Daily (Suspension and Tablet) in the Age Group 12-<18 Years
Description: The aPTT is a screening test for the intrinsic pathway and is sensitive for deficiencies of Factors I, II, V,VIII, IX, X, XI and XII. The initial read-out is in seconds.
Time Frame: Up to 4 hours post dose on Day 30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 12-<18
Number analyzed (Participants) | 154
ratio
  Day 30 (0.5-1.5h) n=154 | 1.17 (0.28)
  Day 30 (2.5-4h) n=149: number analyzed (Participants) | 149
  Day 30 (2.5-4h) n=149 | 1.38 (0.50)
  Day 60 (2-8h) n=153: number analyzed (Participants) | 153
  Day 60 (2-8h) n=153 | 1.33 (0.38)

21. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Ratios to Baseline: Rivaroxaban Administered Once Daily (Suspension and Tablet) in the Age Group 6-<12 Years
Description: as for outcome 20
Time Frame: Up to 4 hours post dose on Day 30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 6-<12
Number analyzed (Participants) | 19
ratio
  Day 30 (0.5-1.5h) n=17: number analyzed (Participants) | 17
  Day 30 (0.5-1.5h) n=17 | 1.27 (0.20)
  Day 30 (2.5-4h) n=17: number analyzed (Participants) | 17
  Day 30 (2.5-4h) n=17 | 1.39 (0.26)
  Day 60 (2-8h) n=19 | 1.24 (0.20)

22. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Ratios to Baseline: Rivaroxaban Administered Twice Daily (Suspension and Tablet) in the Age Group 6-<12 Years
Description: as for outcome 20
Time Frame: Up to 4 hours post dose on Day 30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 6-<12
Number analyzed (Participants) | 31
ratio
  Day 30 (0.5-1.5h) n=30: number analyzed (Participants) | 30
  Day 30 (0.5-1.5h) n=30 | 1.11 (0.24)
  Day 30 (2.5-4h) n=30: number analyzed (Participants) | 30
  Day 30 (2.5-4h) n=30 | 1.15 (0.22)
  Day 60 (2-8h) n=31 | 1.18 (0.24)

23. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Ratios to Baseline: Rivaroxaban Administered Twice Daily (Suspension) in the Age Group 2-<6 Years
Description: The aPTT is a screening test for the intrinsic pathway and is sensitive for deficiencies of Factors I, II, V,VIII, IX, X, XI and XII. The initial read-out is in seconds. 'NA' denotes the data that cannot be calculated.
Time Frame: Up to 4 hours post dose on Day 30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 2-<6
Number analyzed (Participants) | 32
ratio
  Day 30 (0.5-1.5h) n=1: number analyzed (Participants) | 1
  Day 30 (0.5-1.5h) n=1 | 0.90 (NA) — 'NA' denotes data that cannot be calculated.
  Day 30 (2.5-4h) n=32 | 1.29 (0.33)
  Day 60 (2-8h) n=29: number analyzed (Participants) | 29
  Day 60 (2-8h) n=29 | 1.23 (0.21)

24. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Ratios to Baseline: Rivaroxaban Administered Twice Daily (Suspension) in the Age Group 0.5-<2 Years
Description: as for outcome 23
Time Frame: Up to 4 hours post dose on Day 30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 0.5-<2
Number analyzed (Participants) | 2
ratio
  Day 30 (0.5-1.5h) n=0: number analyzed (Participants) | 0
  Day 30 (2.5-4h) n=1: number analyzed (Participants) | 1
  Day 30 (2.5-4h) n=1 | 1.13 (NA) — 'NA' denotes data that cannot be calculated.
  Day 60 (2-8h) n=2 | 1.10 (0.02)

25. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Ratios to Baseline: Rivaroxaban Administered Three Times Daily (Suspension) in the Age Group 2-<6 Years
Description: as for outcome 20
Time Frame: Up to 3 hours post dose on Day 30, and up to 6 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 2-<6
Number analyzed (Participants) | 4
ratio
  Day 30 (0.5-3h) n=4 | 1.50 (0.83) [lower limit 0.83]
  Day 60 (2-6h) n=4 | 1.13 (0.06) [lower limit 0.06]

26. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Ratios to Baseline: Rivaroxaban Administered Three Times Daily (Suspension) in the Age Group 0.5-<2 Years
Description: as for outcome 20
Time Frame: Up to 3 hours post dose on Day 30, and up to 6 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged 0.5-<2
Number analyzed (Participants) | 9
ratio
  Day 30 (0.5-3h) n=9 | 1.20 (0.39)
  Day 60 (2-6h) n=6: number analyzed (Participants) | 6
  Day 60 (2-6h) n=6 | 1.10 (0.47)

27. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Ratios to Baseline: Rivaroxaban Administered Three Times Daily (Suspension) in the Age Group Birth-<0.5 Years
Description: as for outcome 20
Time Frame: Up to 3 hours post dose on Day 30, and up to 6 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rivaroxaban, Aged Birth-<0.5
Number analyzed (Participants) | 9
ratio
  Day 30 (0.5-3h) n=9 | 1.31 (0.15)
  Day 60 (2-6h) n=3: number analyzed (Participants) | 3
  Day 60 (2-6h) n=3 | 1.21 (0.16)

28. Secondary Outcome: Anti-Xa Values: Rivaroxaban Administered Once Daily (Suspension and Tablet) in the Age Group 12-<18 Years
Description: This is a method for measuring the inhibition of Factor Xa activity determined by an ex vivo using a photometric method.
Time Frame: Up to 4 hours post dose on Day 30, up to 8 hours post dose on Day 60, and up to 24 hours on Day 90
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Aged 12-<18
Number analyzed (Participants) | 167
microgram per liter (mcg/L)
  Day 30 (0.5-1.5h) n=141: number analyzed (Participants) | 141
  Day 30 (0.5-1.5h) n=141 | 164.46 (124.46)
  Day 30 (2.5-4h) n=164: number analyzed (Participants) | 164
  Day 30 (2.5-4h) n=164 | 254.66 (188.64)
  Day 60 (2-8h) n=167 | 255.40 (171.59)
  Day 90 (20-24h) n=58: number analyzed (Participants) | 58
  Day 90 (20-24h) n=58 | 62.12 (175.87)

29. Secondary Outcome: Anti-Xa Values: Rivaroxaban Administered Once Daily (Suspension and Tablet) in the Age Group 6-<12 Years
Description: This is a method for measuring the inhibition of Factor Xa activity determined by an ex vivo using a photometric method.
Time Frame: Up to 4 hours post dose on Day 30, up to 8 hours post dose on Day 60, and up to 24 hours on Day 90
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Aged 6-<12
Number analyzed (Participants) | 23
microgram per liter (mcg/L)
  Day 30 (0.5-1.5h) n=22: number analyzed (Participants) | 22
  Day 30 (0.5-1.5h) n=22 | 206.89 (105.01)
  Day 30 (2.5-4h) n=23 | 263.24 (156.73)
  Day 60 (2-8h) n=22: number analyzed (Participants) | 22
  Day 60 (2-8h) n=22 | 243.45 (124.92)
  Day 90 (20-24h) n=9: number analyzed (Participants) | 9
  Day 90 (20-24h) n=9 | 27.39 (14.66)

30. Secondary Outcome: Anti-Xa Values: Rivaroxaban Administered Twice Daily (Suspension and Tablet) in the Age Group 6-<12 Years
Description: This is a method for measuring the inhibition of Factor Xa activity determined by an ex vivo using a photometric method.
Time Frame: Up to 4 hours post dose on Day 30, up to 8 hours post dose on Day 60, and up to 16 hours on Day 90
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Aged 6-<12
Number analyzed (Participants) | 37
microgram per liter (mcg/L)
  Day 30 (0.5-1.5h) n=37 | 96.82 (76.77)
  Day 30 (2.5-4h) n=36: number analyzed (Participants) | 36
  Day 30 (2.5-4h) n=36 | 139.10 (102.19)
  Day 60 (2-8h) n=35: number analyzed (Participants) | 35
  Day 60 (2-8h) n=35 | 126.53 (81.78)
  Day 90 (10-16h) n=20: number analyzed (Participants) | 20
  Day 90 (10-16h) n=20 | 47.49 (66.88)

31. Secondary Outcome: Anti-Xa Values: Rivaroxaban Administered Twice Daily (Suspension) in the Age Group 2-<6 Years
Description: This is a method for measuring the inhibition of Factor Xa activity determined by an ex vivo using a photometric method.
Time Frame: Up to 4 hours post dose on Day 30, up to 8 hours post dose on Day 60, and up to 16 hours on Day 90
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Aged 2-<6
Number analyzed (Participants) | 37
microgram per liter (mcg/L)
  Day 30 (2.5-4h) n=37 | 177.78 (147.29)
  Day 60 (2-8h) n=36: number analyzed (Participants) | 36
  Day 60 (2-8h) n=36 | 150.03 (95.77)
  Day 90 (10-16h) n=18: number analyzed (Participants) | 18
  Day 90 (10-16h) n=18 | 54.40 (51.52)

32. Secondary Outcome: Anti-Xa Values: Rivaroxaban Administered Twice Daily (Suspension) in the Age Group 0.5-<2 Years
Description: This is a method for measuring the inhibition of Factor Xa activity determined by an ex vivo using a photometric method. 'NA' denotes the data that cannot be calculated.
Time Frame: Up to 4 hours post dose on Day 30, and up to 8 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Aged 0.5-<2
Number analyzed (Participants) | 4
microgram per liter (mcg/L)
  Day 30 (0.5-1.5h) n=1: number analyzed (Participants) | 1
  Day 30 (0.5-1.5h) n=1 | 247.54 (NA) — 'NA' denotes data that cannot be calculated.
  Day 30 (2.5-4h) n=2: number analyzed (Participants) | 2
  Day 30 (2.5-4h) n=2 | 160.71 (153.84)
  Day 60 (2-8h) n=4 | 121.09 (81.94)

33. Secondary Outcome: Anti-Xa Values: Rivaroxaban Administered Three Times Daily (Suspension) in the Age Group 2-<6 Years
Description: as for outcome 32
Time Frame: Up to 3 hours post dose on Day 30, up to 6 hours post dose on Day 60, and up to 16 hours on Day 90
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Aged 2-<6
Number analyzed (Participants) | 4
microgram per liter (mcg/L)
  Day 30 (0.5-3h) n=4 | 209.67 (127.86)
  Day 60 (2-6h) n=4 | 140.46 (78.82)
  Day 90 (10-16h) n=1: number analyzed (Participants) | 1
  Day 90 (10-16h) n=1 | 62.56 (NA) — 'NA' denotes data that cannot be calculated.

34. Secondary Outcome: Anti-Xa Values: Rivaroxaban Administered Three Times Daily (Suspension) in the Age Group 0.5-<2 Years
Description: as for outcome 32
Time Frame: Up to 3 hours post dose on Day 30, up to 6 hours post dose on Day 60, up to 16 hours on Day 90 and follow-up up to 30 days
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Aged 0.5-<2
Number analyzed (Participants) | 12
microgram per liter (mcg/L)
  Day 30 (0.5-3h) n=12 | 111.35 (97.03)
  Day 30 (2-6h) n=11: number analyzed (Participants) | 11
  Day 30 (2-6h) n=11 | 147.24 (125.40)
  Day 90 (10-16h) n=3: number analyzed (Participants) | 3
  Day 90 (10-16h) n=3 | 23.40 (4.51)
  Follow-up n=1: number analyzed (Participants) | 1
  Follow-up n=1 | 71.30 (NA) — 'NA' denotes data that cannot be calculated.

35. Secondary Outcome: Anti-Xa Values: Rivaroxaban Administered Three Times Daily (Suspension) in the Age Group Birth-<0.5 Years
Description: This is a method for measuring the inhibition of Factor Xa activity determined by an ex vivo using a photometric method.
Time Frame: Up to 3 hours post dose on Day 30, and up to 6 hours post dose on Day 60
Population: Participants in pharmacodynamics set (PDS) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Aged Birth-<0.5
Number analyzed (Participants) | 10
microgram per liter (mcg/L)
  Day 30 (0.5-3h) n=10 | 118.12 (82.08)
  Day 60 (2-6h) n=5: number analyzed (Participants) | 5
  Day 60 (2-6h) n=5 | 228.03 (181.08)

ADVERSE EVENTS:
Time Frame: After randomization until last intake of study medication plus 2 days, up to 1 year
Arm/Group | Comparator Group | Rivaroxaban Group
All-Cause Mortality (participants affected / at risk) | 0/162 | 2/329
Serious Adverse Events (participants affected / at risk) | 35/162 | 78/329
Other Adverse Events (participants affected / at risk) | 121/162 | 275/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comparator Group (N=162) | Rivaroxaban Group (N=329)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 8 (9)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Muscular dystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (6)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 2 (3) | 6 (6)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2)
Eczema herpeticum (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (3)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pyoderma streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental underdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incorrect route of product administration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Drug clearance decreased (Investigations) | 1 (1) | 0 (0)
Gastrointestinal stoma output decreased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (2)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Sciatic nerve neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 1 (2) | 0 (0)
Hemianaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Colostomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Mastoidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Sclerotherapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Lumboperitoneal shunt (Surgical and medical procedures) | 0 (0) | 1 (1)
Faecal disimpaction (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comparator Group (N=162) | Rivaroxaban Group (N=329)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 11 (20)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (8)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (5)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 6 (7)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 10 (15)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (2) | 1 (2)
Autoimmune neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 6 (6)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Immunodeficiency congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Protein S deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 6 (7)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0)
Amblyopia (Eye disorders) | 0 (0) | 1 (1)
Astigmatism (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 2 (2)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Heterophoria (Eye disorders) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 2 (2)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1)
Optic disc haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Papilloedema (Eye disorders) | 3 (3) | 4 (5)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 2 (2)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 17 (27)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 11 (12)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (4)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (10) | 8 (11)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 25 (30)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 13 (13)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 6 (6)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (7) | 22 (25)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 7 (8)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 4 (7)
Tongue blistering (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 3 (4)
Vomiting (Gastrointestinal disorders) | 13 (17) | 36 (42)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 1 (2)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (2)
Asthenia (General disorders) | 1 (1) | 3 (5)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 5 (6) | 16 (18)
Cyst (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (6) | 21 (23)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Granuloma (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 2 (2)
Injection site bruising (General disorders) | 8 (8) | 0 (0)
Injection site extravasation (General disorders) | 1 (2) | 0 (0)
Injection site haematoma (General disorders) | 3 (3) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 1 (3) | 0 (0)
Injection site mass (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 4 (4)
Oedema (General disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 4 (4)
Pain (General disorders) | 0 (0) | 7 (7)
Pyrexia (General disorders) | 14 (22) | 37 (51)
Application site vesicles (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 4 (5) | 5 (5)
Catheter site haemorrhage (General disorders) | 1 (1) | 1 (1)
Puncture site haemorrhage (General disorders) | 5 (8) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Catheter site rash (General disorders) | 1 (1) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Application site hypersensitivity (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 0 (0)
Medical device site haemorrhage (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (2) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Secondary immunodeficiency (Immune system disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2) | 3 (4)
Ear infection (Infections and infestations) | 1 (1) | 3 (3)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 7 (7)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 4 (4)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (4) | 6 (6)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 3 (4)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (13) | 29 (36)
Oral candidiasis (Infections and infestations) | 1 (1) | 5 (5)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 3 (3)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 3 (3)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (3) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 4 (4) | 11 (12)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 6 (6)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 4 (4) | 5 (5)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 10 (13)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 4 (4)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Oral infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 2 (2)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (2)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Mastoid abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection viral (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 4 (5)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 7 (7)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 5 (6)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Greenstick fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (4)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 5 (5) | 14 (21)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 9 (10) | 15 (19)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Wound haemorrhage (Injury, poisoning and procedural complications) | 2 (3) | 13 (14)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Underdose (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site rash (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental underdose (Injury, poisoning and procedural complications) | 0 (0) | 7 (8)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebral radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Product prescribing error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase abnormal (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (10) | 6 (11)
Aspartate aminotransferase abnormal (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 6 (10)
Aspiration bone marrow (Investigations) | 0 (0) | 1 (2)
Bilirubin conjugated increased (Investigations) | 0 (0) | 3 (4)
Biopsy liver (Investigations) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 4 (4)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Coagulation factor VIII level increased (Investigations) | 2 (2) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 2 (2)
Full blood count abnormal (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 3 (3)
International normalised ratio abnormal (Investigations) | 1 (1) | 0 (0)
Lumbar puncture (Investigations) | 0 (0) | 1 (3)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (4)
Neutrophil count increased (Investigations) | 0 (0) | 1 (2)
Nuclear magnetic resonance imaging (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 9 (20)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 3 (3)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte percentage decreased (Investigations) | 0 (0) | 1 (1)
Lipoprotein (a) increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 1 (2)
Blood alkaline phosphatase decreased (Investigations) | 0 (0) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 3 (3)
Angiogram (Investigations) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Epstein-Barr virus test positive (Investigations) | 0 (0) | 1 (1)
Clostridium test positive (Investigations) | 0 (0) | 1 (1)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1)
Chlamydia test positive (Investigations) | 0 (0) | 1 (1)
Influenza B virus test positive (Investigations) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Human rhinovirus test positive (Investigations) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 8 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Selenium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 12 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (12) | 23 (25)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Clumsiness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 11 (11)
Dizziness exertional (Nervous system disorders) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 24 (28) | 56 (75)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 2 (2)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 5 (5)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
VIth nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Toxic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Choroid fissure cyst (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (5)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Mood altered (Psychiatric disorders) | 2 (2) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Somnambulism (Psychiatric disorders) | 0 (0) | 1 (1)
Phonophobia (Psychiatric disorders) | 0 (0) | 1 (1)
Post stroke depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 5 (8)
Hypercalciuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal atrophy (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 4 (5)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (3) | 2 (2)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 4 (11)
Genital rash (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 5 (6) | 21 (29)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Polycystic ovaries (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 4 (10)
Genital tract inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Perineal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 18 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 (32) | 40 (62)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (7)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural adhesion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 13 (16)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (9)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (8)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 17 (19)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Bladder catheterisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Intra-uterine contraceptive device insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Ventricular drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrointestinal tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 3 (3)
Hepatitis B immunisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Oophorectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Mastoid operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 4 (5)
Stem cell transplant (Surgical and medical procedures) | 0 (0) | 1 (2)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Endotracheal intubation (Surgical and medical procedures) | 0 (0) | 1 (1)
Ventriculo-cardiac shunt (Surgical and medical procedures) | 0 (0) | 1 (1)
Laryngeal mask airway insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 2 (5)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 3 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Superficial vein prominence (Vascular disorders) | 1 (1) | 0 (0)
May-Thurner syndrome (Vascular disorders) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT02234843/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT02234843/SAP_001.pdf